CLINICAL TRIAL: NCT04061993
Title: Effects of Early Home-based Strength and Sensory-motor Training After Total Hip Arthroplasty: a Randomised Controlled Trial
Brief Title: Effects of Early Home-based Strength and Sensory-motor Training After THA on Functional Outcome and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valdoltra Orthopedic Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PRT_PhD
Record Dates: First submitted 2019-07-11; First posted 2019-08-20 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Arthroplasty; Replacement; Hip; Strength Training
Keywords: Total hip arthroplasty; Early postoperative exercise; Home-based training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention Group OBV (Experimental): Intervention Group in Valdoltra Orthopaedic Hospital. Patients will get current standard physiotherapy during hospitalisation and extra one-on-one training to learn strength and sensory-motor exercises. At discharge they will get USB drives with exercise videos, written exercise instructions, training diary and exercise aids for strength and sensory-motor training.
  Interventions: Procedure: Strength and Sensory-Motor Training; Procedure: Current Standard Physiotherapy
- Control Group OBV (Active Comparator): Control Group in Valdoltra Orthopaedic Hospital. Patients will get current standard physiotherapy during hospitalisation and USB drives with exercise videos, written exercise instructions and training diary at discharge.
  Interventions: Procedure: Current Standard Physiotherapy
- Intervention Group SBNM (Experimental): Intervention Group in General Hospital Novo mesto. Patients will get current standard physiotherapy during hospitalisation and extra one-on-one training to learn strength and sensory-motor exercises. At discharge they will get USB drives with exercise videos, written exercise instructions, training diary and exercise aids for strength and sensory-motor training.
  Interventions: Procedure: Strength and Sensory-Motor Training; Procedure: Current Standard Physiotherapy
- Control Group SBNM (Active Comparator): Control Group in General Hospital Novo mesto. Patients will get current standard physiotherapy during hospitalisation and USB drives with exercise videos, written exercise instructions and training diary at discharge.
  Interventions: Procedure: Current Standard Physiotherapy

INTERVENTIONS:
Procedure: Strength and Sensory-Motor Training — Early postoperative strength and sensory-motor training after total hip arthroplasty. Training consists of: hip muscles strengthening (focusing on abductors); hip and pelvic stabilization exercises; ankle and knee muscles strengthening (better dissipation of impact forces and femoral inner rotation control); trunk muscles strengthening (stabilization of pelvis and lumbar spine and reduction of local loading).
  Arms: Intervention Group OBV; Intervention Group SBNM
Procedure: Current Standard Physiotherapy — Mobilisation using a walking aid (usually two crutches, rarely a walker), deep vein thrombosis (DVT) prevention exercises, lower limb range of motion exercises and isometric strengthening program

SUMMARY:
A prospective multicentre randomised clinical trial of 250 selected patients with THA, who will be randomly assigned to intervention (IG) or control group (CG). Both will have standard physiotherapy during hospitalisation, IG will additionally learn strength and sensory-motor training exercises. Follow up will be performed with physical tests, maximal voluntary isometric contractions and outcome assessment questionnaires at baseline and 1, 3 and 12 months after surgery.

DETAILED DESCRIPTION:
This study is a prospective multicentre randomised clinical trial to be conducted in orthopaedic departments of two Slovenian hospitals. In each hospital 125 patients aged 60 or older with unilateral osteoarthritis, ASA score 1-3, signed informed consent, access to watching USB videos and without terminal illnesses disabling rehabilitation participation, will be randomly assigned to intervention (IG) or control group (CG). Total hip arthroplasty with anterior approach will be performed. All patients will get current standard physiotherapy during hospitalisation. Patients in IG will additionally learn strength and sensory-motor training exercises. Patients in both groups will get USB drives with exercise videos, written exercise instructions and training diary. Physiotherapists will perform measurements (physical tests and maximal voluntary isometric contractions) and patients will fill in outcome assessment questionnaires (Harris Hip Score and 36-Item Short Form Health Survey) at baseline and 1, 3 and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective primary unilateral THA for OA.
2. Patients older than 60 years at the time of surgery.
3. Ability to watch exercise videos on USB drive.
4. American Society of Anaesthesiologists (ASA) Classification 1-3.
5. Patients are able to consent and willing to comply with the study protocol.

Exclusion Criteria:

1. Primary THA for a diagnosis other than OA (aseptic femoral head necrosis, dysplastic hip…) or revision THA.
2. Patients having previous hip interventions (osteosynthesis, osteotomy…)
3. Discharge to rehabilitation units or nursing homes.
4. Patients unable to consent and comply with the study protocol (diagnosed with dementia, mental disorders, poor preoperative physical status - neurological disorders, amputations, trouble walking with walkers or wheelchairs, painful hip or knee prosthesis in other joints).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Change in isometric hip and trunk muscles strength | Baseline (before surgery), 1, 3 and 12 months after surgery
  Maximal voluntary isometric contractions. We will use specially prepared measuring device with dynamometer attached to stiff bands metal chains. For the assessment of maximal isometric strength, a maximal voluntary isometric contraction for 6 seconds is asked. The same procedure to obtain a maximal voluntary contraction is used for every strength measure. 3 movement planes are assessed for trunk (extension, left and right abduction) and operated hip (flexion, extension and abduction) and 2 for opposite hip (extension, abduction).
Change in 8UG | Baseline (before surgery), 1, 3 and 12 months after surgery
  8-Feet Up and Go Test. The 8UG is a timed test that requires one to stand up from a chair with armrests, walk to a cone 8 feet away, turn around, return to the chair and sit down.
Change in 10MW | Baseline (before surgery), 1, 3 and 12 months after surgery
  Timed 10-meter walk test. Individual walks without assistance 10 meters and the time is measured for the intermediate 6 meters to allow for acceleration and deceleration. The test is first performed at preferred walking speed and second at fastest speed possible.

SECONDARY OUTCOMES:
HHS | Baseline (before surgery), 1, 3 and 12 months after surgery
  Harris Hip Score. The HHS is a widely used disease-specific measure of hip disabilities after THA. The physiotherapist administers the test in the form of a structured interview with the patients. The domains include pain, functions of daily living and gait. The rating scale is from 0 (worse) to 100 points (best). The HHS is considered to have good validity and reliability.
SF-36_v2 | Baseline (before surgery), 3 and 12 months after surgery
  36-item short form health survey. The SF-36v2 is a multipurpose, short-form 36-item health survey yielding a profile of two health component summary measures: psychometrically-based physical component summary (PCS) and mental component summary (MCS) scores. It consists of eight health domain scales: Physical functioning (PF), Role-Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role-Emotional (RE) and Mental Health (MH). The interpretation of results in simplified with the norm-based scoring (Mean = 50, SD = 10) of its health domain scales and component summary measures.

OTHER OUTCOMES:
Training compliance | First 3 months after surgery
  Training dairy. All participants in both groups will keep a training dairy concerning all training activities - they will make marks by every exercise they will perform on exact day, write notes if they will have any other sport activities (walking, stationary bicycling and other) and if there will be any adverse effects, reasons why they skipped training if they did. They will also measure pain on Visual Analog Scale (VAS) during day before and after training and during night.

CONTACTS AND LOCATIONS:
Locations (2):
- Slovenia (2):
  - Valdoltra Orthopaedic Hospital, Ankaran
  - General Hospital Novo mesto, Novo Mesto

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and analysed during the current study are and will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Kristof Mirt P, Strojnik V, Kavcic G, Trebse R. Effects of early home-based strength and sensory-motor training after total hip arthroplasty: study protocol for a multicenter randomized controlled trial. Trials. 2022 Nov 8;23(1):929. doi: 10.1186/s13063-022-06779-8. PMID 36348372